CLINICAL TRIAL: NCT03394573
Title: A Randomized, Study Investigating the Efficacy of Visual Acuity-based Versus Optical Coherence Tomography (OCT) -Based Treat and Extend Regimen Using Aflibercept in Patients With Diabetic Macular Edema
Brief Title: Comparison of VA Guided Versus OCT Guided TER Using Aflibercept for Diabetic Macular Edema (AVOCT Study)
Acronym: AVOCT
Status: Terminated | Type: Observational
Why Stopped: insufficient recuritment due to covid
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: AVOCT
Record Dates: First submitted 2016-01-04; First posted 2018-01-09 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic macular edema
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- OCT guided treatment arm: OCT guided aflibercept injection
  Interventions: Other: OCT guided treatment arm
- VA guided treatment arm: VA guided aflibercept injection
  Interventions: Other: VA guided treatment arm

INTERVENTIONS:
Other: OCT guided treatment arm — Intravitreal injection of Aflibercept for DME OCT guided
  Other Names: aflibercept
  Groups: OCT guided treatment arm
Other: VA guided treatment arm — Intravitreal injection of Aflibercept for DME VA guided
  Other Names: aflibercept
  Groups: VA guided treatment arm

SUMMARY:
This study will evaluate the effectiveness of aflibercept (Eylea®) using two different treatment protocols in patients with vision loss from diabetic macular edema. While one group will be treated with an optical coherence tomography (OCT) guided 'treat and extend' regimen, the other group will be treated according to a visual acuity (VA) guided 'treat and extend' protocol. The patients will be randomized into two treatment arms using an automated randomization algorithm.

DETAILED DESCRIPTION:
For the study arm receiving the VA-guided treatment regimen, the following retreatment criteria will be applied:

* if visual acuity remains stable (± 5 ETDRS letters) treatment intervals will be extended by 2 weeks as compared to the previous retreatment interval.
* if visual acuity decreases by more than 5 ETDRS letters treatment intervals will be shortened by 1 week as compared to the previous retreatment interval, whereby retreatment intervals cannot be shorter than 28 days (4 weeks). Once treatment intervals have been shortened, the patient should be seen at two consecutive visits with no diabetic retinopathy disease activity before re-extending the treatment interval.

For the study arm receiving the OCT-guided treatment regimen, the following retreatment criteria will be applied:

* if SD-OCT examinations show 1) no SRF in any area of the OCT scan present and 2) no IRF, treatment intervals will be extended by 2 weeks as compared to the previous retreatment interval.
* if SD-OCT examinations show 1) any SRF present in any area of the OCT scan and/or 2) any IRF present, treatment intervals will be shortened by 1 week as compared to the previous retreatment interval, whereby retreatment intervals cannot be shorter than 28 days (4 weeks). Once treatment intervals have been shortened, the patient should be seen at two consecutive visits with no diabetic retinopathy disease activity before re-extending the treatment interval.

ELIGIBILITY:
General:

* Informed consent as documented by signature of the patient on the informed consent form.
* Male or female, ≥ 18 years of age.
* Patients with Type 1 or Type 2 diabetes mellitus (according to ADA or WHO guidelines).
* No relevant change in medication for the management of diabetes within 3 months prior to randomization.
* Patients fulfilling criteria specified in the respective SmPC for aflibercept for the treatment of DME

Study eye:

* Visual impairment due to focal or diffuse DME in at least one eye. If both eyes are eligible, the eye with the worse visual acuity, as assessed at Visit 1, will be selected for study treatment unless, based on medical reasons, the investigator deems the other eye the more appropriate candidate for study treatment.
* BCVA score between 78 and 39 letters using ETDRS- visual acuity testing charts at a testing distance of 4 meters (approximate Snellen equivalent of 20/32 to 20/160) Decrease in vision and CRT due to DME and not due to other causes, at the investigators discretion

Inclusion criteria:

General:

* Informed consent as documented by signature of the patient on the informed consent form.
* Male or female, ≥ 18 years of age.
* Patients with Type 1 or Type 2 diabetes mellitus (according to ADA or WHO guidelines).
* No relevant change in medication for the management of diabetes within 3 months prior to randomization.
* Patients fulfilling criteria specified in the respective SmPC for aflibercept for the treatment of DME

Study eye:

* Visual impairment due to focal or diffuse DME in at least one eye. If both eyes are eligible, the eye with the worse visual acuity, as assessed at Visit 1, will be selected for study treatment unless, based on medical reasons, the investigator deems the other eye the more appropriate candidate for study treatment.
* BCVA score between 78 and 39 letters using ETDRS- visual acuity testing charts at a testing distance of 4 meters (approximate Snellen equivalent of 20/32 to 20/160) Decrease in vision and CRT due to DME and not due to other causes, at the investigators discretion

Exclusion criteria:

General:

* Inability to comply with study or follow-up procedures.
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential, not using or not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the Investigator in individual cases.(Female participants who are surgically sterilised/ hysterectomised, or post-menopausal for longer than 2 years are not considered as being of child-bearing potential.)
* Any type of systemic disease or its treatment, in the opinion of the Investigator, including any medical condition (controlled or uncontrolled) that could be expected to progress, recur, or change to such an extent that it may bias the assessment of the clinical status of the patient to a significant degree.
* Stroke or myocardial infarction less than 3 months prior to the date of informed consent signature.
* Known hypersensitivity to aflibercept or any component of the aflibercept formulation. Any other reason that would prevent treatment with aflibercept specified in the SmPC
* Current use of any systemic anti- VEGF drugs [e.g., bevacizumab (Avastin®)].
* Use of other investigational drugs at screening visit.

Both eyes:

* Any active ocular infection or inflammation (scleritis, uveitis, endophthalmitis) at the time of screening or baseline.
* Uncontrolled glaucoma [intraocular pressure (IOP) ≥30 mmHg on medication or according to Investigator's judgment] at the time of screening or baseline.
* Neovascularisation of the iris or neovascular glaucoma at the time of screening or baseline.
* Intravitreal corticosteroids administered within 3 months prior to the date of informed consent signature.

Study eye:

* Visually significant cataract, vitreous hemorrhage, rhegmatogenous retinal detachment or age related macular degeneration
* Intraocular treatment with any anti-VEGF drug or intravitreal corticosteroids prior to the date of informed consent signature.
* Inability of obtaining SD-OCT images of sufficient quality to be analysed
* Any intraocular procedure anticipated within the next 6 months following the date of informed consent signature

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with vision loss due to diabetic macular edema
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2017-09-16 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Functional outcomes | 24 months
  Mean change in BCVA from baseline to week 104 (EOS)

SECONDARY OUTCOMES:
Number of visits | 24 months
  Number of visits per Treatment arm
Number of injections | 24 months
  Number of injections per Treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Martin Zinkernagel, MD, PhD, Study Director — University of Bern, Switzerland; Marion Munk, MD, PhD, Principal Investigator — University of Bern, Switzerland
Locations (1):
- Inselspital Bern, Department of Ophthalmology, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No